CLINICAL TRIAL: NCT03339583
Title: Effectiveness of Nonspecific Methods of Treatment and Zopiclone for Chronic Insomnia
Brief Title: Effectiveness of BBT-I and Zopiclone for Chronic Insomnia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Polina Pchelina, Postgraduate student. Institute of Professional Education, Chair of Neurology. I.M. Sechenov First Moscow State Medical University, I.M. Sechenov First Moscow State Medical University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2017-10-17; First posted 2017-11-13 (Actual); Results first posted 2019-06-17 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Insomnia Chronic
Keywords: chronic insomnia; brief behavioral treatment; behavioral treatment; insomnia severity index; predictors; treatment response
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — zopiclone; Hypnotics and Sedatives

STUDY DESIGN:
Intervention Model Description: Study design implied that every patient underwent two different treatment courses in random sequence: hypnotic or structured educational program (BBT-I) delivered in two sessions.
  Subjects were randomly assigned to one of treatment sequences by card sorting method. Patients of the zopiclone-first group underwent the medication therapy for the first two weeks followed by educational program. Patients of the BBT-I-first group received two-week educational program followed by medication therapy.
  Each treatment course was separated by 2-weeks washout period that provided the opportunity to evaluate the sustainability of treatment effect.
  Before and after each treatment course and after each washout period subjects completed set of questionnaires.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- zopiclone first group (Experimental): underwent the medication therapy (zopiclone) for the first two weeks followed by brief behavioral therapy
  Interventions: Behavioral: Brief behavioral therapy; Drug: Zopiclone
- BBT-I first group (Experimental): received two-week brief behavioral therapy followed by medication therapy (zopiclone).
  Interventions: Behavioral: Brief behavioral therapy; Drug: Zopiclone

INTERVENTIONS:
Behavioral: Brief behavioral therapy — program included a question-and-answer part; a didactic presentation of sleep regulation mechanisms; the review of causes of onset and chronification of illness; an examination of patient's sleep log; explanation of sleep restriction method and prescription of individual regimen of sleep; explanation of stimulus control method; sleep hygiene education; discussion of relaxation techniques. Participants were supplied with 32 minute audio recording "Relaxation and refreshment session for insomnia" created for this study by Dr. A.Tabidze with verbal relaxing instructions with quiet musical composition behind it. Participants were instructed to listen to this recording in headphones each day for 2-week BBT-I period after laying into bed and turning the light off.
  Other Names: BBT-I
Drug: Zopiclone — zopiclone intake in a dose of 7,5 mg 30 minutes before bedtime for two weeks
  Other Names: hypnotic

SUMMARY:
Background: Importance of chronic insomnia (CI) problem is determined by its high prevalence rate, comorbidity and resistance to the treatment. Although cognitive behavior treatment of insomnia (CBT-I) remains the recommended treatment for CI it has disadvantages of time consuming and low treatment response. Hence shortened and simplified behavioral approaches such as Brief Behavioral therapy of insomnia (BBT-I) are developed. The aim of the present study is to test the effectiveness of BBT-I program for chronic insomnia in comparison with zopiclone in Russian population. The anthropometric, psychological and polysomnographic characteristics of patients were measured to find predictors of effectiveness of each method.

Participants: 42 adults (14 males, 28 females, mean age 54 years) meeting the criteria for CI according International classification of sleep disorders-3 Methods: Participants were randomized into two groups. Each group passed 2-week courses of treatment by brief behavior treatment of insomnia (BBT-I) and zopiclone in different orders with 2-week washout period between the courses. Participants underwent in-lab polysomnography prior to the treatment and completed questionnaires (Insomnia Severity Index (ISI), Dysfunctional beliefs about sleep scale (DBAS), Beck Depression Inventory (BDI) and others) in the beginning and the end of each course

DETAILED DESCRIPTION:
The study had a crossover design implying that every patient underwent two different treatment courses in random sequence: hypnotic or structured educational program (BBT-I) delivered in two sessions.

Each treatment course was separated by 2-weeks washout period that provided the opportunity to evaluate the sustainability of treatment effect.

Before and after each treatment course and after each washout period subjects completed set of questionnaires.

The total duration of the study was 8 weeks in which 6 visits including 1 night polysomnography (PSG), 2 face-to-face structured educational program sessions and 5 diagnostic interviews have been performed.

Participants A sample of 42 adults (14 males, 28 females, mean age 54 years from 29 to 80 years) meeting the criteria for chronic insomnia according ICSD-3 was recruited from outpatient care of Department of sleep medicine of University Hospital №3 of I.M. Sechenov First Moscow State Medical University. All participants were informed about the nature, purpose, risks, and discomforts that could arise from their participation, and about their right to withdraw at any time. Subjects documented their willingness to participate by signing the informed consent form, approved by local Ethic Committee.

Treatment methods. BBT-I program includes two weekly one hour individual sessions; Hypnotic (zopiclone) in a dose of 7,5 mg has to be taken 30 minutes before bedtime for two weeks

Measures Questionnaires. During the first visit patients underwent structured clinical interview and filled in self-report questionnaires: Beck Depression Inventory (BDI), State-trait anxiety inventory (STAI), Toronto Alexithymia Scale - short version (TAS-20) , Big Five Questionnaire (BFQ-2R), Pittsburgh Sleep Quality Index (PSQI), Insomnia Severity Index (ISI), Dysfunctional beliefs about sleep scale (DBAS), Sleep hygiene index (SHI).

During the next 4 visits participants repeatedly underwent diagnostic tests included BDI, STAI, PSQI, ISI, DBAS, SHI.

Participants kept daily sleep diaries where they recorded bedtime and morning rise time, sleep onset latency (SOL), number of night awakenings and time of wakefulness after sleep onset before waking up (WASO) for the whole study period.

On the last visit participants completed questionnaire for assessment of effectiveness of treatment along with diagnostic routine. Patients were asked to rank the effectiveness of proposed methods of treatment (didactic presentation, stimulus control, sleep restriction, relaxing recording and zopiclone) in ascending order from 1 to 5 points (5 seems most effective).

Polysomnography. Participants underwent in-lab PSG (1 night without adaptation night) prior to the treatment in order to exclude other disorders producing subjective sleep complaints (sleep apnea, periodic limb movements disorder). Standard polysomnography montage including 6 monopolar electroencephalography (EEG) channels; 1 submental electromyogram (EMG) channel; 2 electrooculogram (EOG) channels; 2 EMG channels of the right and left tibialis anterior muscles; 1 electrocardiogram channel; oronasal airflow pressure; thoracic and abdominal efforts; respiratory sound; oxygen saturation; body position with videomonitoring was performed. The objective sleep measures included total sleep time (TST), sleep-onset latency, wake time after sleep onset (WASO), number of awakenings, sleep efficiency (the ratio of TST to time spent in bed multiplied on 100%, SE), percentage of sleep stages. PSG data were analysed according the 2007 American Academy of Sleep Medicine criteria including its revision in 2012.

ELIGIBILITY:
Inclusion Criteria:

meeting the criteria for chronic insomnia according ICSD-3 willingness to take part in the study and signed informed consent form

Exclusion Criteria:

1. unability to stop taking medications that have a proven impact on sleep at least one week before and during the study;
2. history of alcohol or drug abuse;
3. major depressive disorder or other severe mental disorder identified by a clinical assessment and medical history;
4. dementia;
5. pregnancy or lactation;
6. shift or night work;
7. medical problems that would be a direct cause of sleep complaints: moderate/severe sleep apnea, defined as an apnea-hypopnea index of ≥15 events per hour, periodic limb movement disorder defined as a periodic leg movement index ≥15 events per hour or restless legs syndrome;
8. other serious chronic conditions or exacerbation of chronic disorder preventing further participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-04-07 (Actual); Primary Completion 2017-03-14 (Actual); Study Completion 2017-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Polina Pchelina, PG student, Principal Investigator — I.M. Sechenov First Moscow State Medical University

IPD SHARING:
Plan to Share IPD: No
Since our lab has no plans to continue or extend the registered study we are not planning share individual patient data with other researches

REFERENCES:
- [Result] Pchelina PV, Tabidze AA, Poluektov MG. [Comparative study of effectiveness of cognitive-behavior therapy and zopiclone for chronic insomnia]. Zh Nevrol Psikhiatr Im S S Korsakova. 2017;117(4. Vyp. 2):48-55. doi: 10.17116/jnevro20171174248-55. Russian. PMID 28777364

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The decision to recruit more patients than it was stated in protocol was made because of dropout of 3 patients and in order to get enough experimental data to provide statistical power
Groups:
- Zopiclone First, Then BBT-I: Participants first received zopiclone in a dose of 7.5 mg 30 minutes before bedtime for two weeks. After a washout of two weeks they then received Brief behavioral therapy program for two weeks in two weekly individual sessions. Then they completed follow-up for two weeks
- BBT-I First, Then Zopiclone: Participants first received Brief behavioral therapy program for two weeks in two weekly individual sessions. After a washout of two weeks they then received zopiclone in a dose of 7.5 mg 30 minutes before bedtime for two weeks. Then they completed follow-up for two weeks
Period: First Intervention (14 Days)
Arm/Group | Zopiclone First, Then BBT-I | BBT-I First, Then Zopiclone
Started | 19 | 23
Completed | 18 | 23
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Washout (14 Days)
Arm/Group | Zopiclone First, Then BBT-I | BBT-I First, Then Zopiclone
Started | 18 | 23
Completed | 18 | 23
Not Completed | 0 | 0
Period: Second Intervention (14 Days)
Arm/Group | Zopiclone First, Then BBT-I | BBT-I First, Then Zopiclone
Started | 18 | 23
Completed | 18 | 21
Not Completed | 0 | 2
Not completed — unrelated acute exacerbation | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Follow-up (14 Days)
Arm/Group | Zopiclone First, Then BBT-I | BBT-I First, Then Zopiclone
Started | 18 | 21
Completed | 12 | 18
Not Completed | 6 | 3
Not completed — Physician Decision | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zopiclone First Group | BBT-I First Group | Total
Number analyzed (Participants) | 19 | 23 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 20 | 33
  >=65 years | 6 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (14.8) | 47.5 (14.1) | 50.7 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 16 | 27
  Male | 8 | 7 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 19 | 23 | 42
Beck depression inventory [Mean (Standard Deviation); unit: units on a scale] — 0-63 scores. higher values represent worse outcome
  units on a scale | 10.8 (5.0) | 12.8 (7.2) | 12.1 (6.1)
State anxiety inventory [Mean (Standard Deviation); unit: units on a scale] — 0-80 scores. higher values represent worse outcome
  units on a scale | 43.5 (8.7) | 46.9 (6.9) | 45.3 (8.1)
trait anxiety inventory [Mean (Standard Deviation); unit: units on a scale] — 0-80 scores. higher values represent worse outcome
  units on a scale | 49.6 (8.3) | 49.1 (7.2) | 49.3 (7.5)
Dysfunctional beliefs about sleep scale [Mean (Standard Deviation); unit: units on a scale] — Measure Description: 0-160 scores. higher values represent worse outcome
  units on a scale | 105.3 (28.7) | 104.9 (30.2) | 105.1 (27.2)
Sleep hygiene index [Mean (Standard Deviation); unit: units on a scale] — Measure Description: 0-65 scores. higher values represent worse outcome
  units on a scale | 26.7 (6.3) | 28.7 (7.3) | 27.9 (6.1)
Insomnia severity index [Mean (Standard Deviation); unit: units on a scale] — 0-28 scores. higher values represent worse outcome
  units on a scale | 18.7 (4.1) | 17.5 (5.4) | 18.6 (4.6)
Pittsburgh sleep quality index [Mean (Standard Deviation); unit: units on a scale] — Measure Description: 0-24 scores. higher values represent worse outcome
  units on a scale | 13.3 (3.5) | 14.5 (2.7) | 14.0 (3.1)
Toronto Alexithymia scale-20 [Mean (Standard Deviation); unit: units on a scale] — Measure Description: 0-100 scores. higher values represent worse outcome
  units on a scale | 49.8 (15.9) | 49.3 (10.0) | 49.5 (12.9)
Sleep efficiency [Mean (Standard Deviation); unit: percentage of polysomnogram time] — derived from 1-night polysomnography at baseline
  percentage of polysomnogram time | 64.68 (17.9) | 63.3 (18.0) | 63.9 (17.7)
sleep latency [Mean (Standard Deviation); unit: minutes] — derived from 1-night polysomnography
  minutes | 38.5 (21.7) | 54.5 (51.0) | 47.0 (40.2)
Wake after sleep onset [Mean (Standard Deviation); unit: minutes] — derived from 1-night polysomnography
  minutes | 102.4 (69.0) | 104.8 (76.1) | 103.6 (71.9)
Awakenings [Mean (Standard Deviation); unit: awakenings] — derived from 1-night polysomnography
  awakenings | 13.8 (6.1) | 13.3 (6.9) | 13.5 (6.5)
N1 NREM sleep percentage [Mean (Standard Deviation); unit: percentage of time] — derived from 1-night polysomnography
  percentage of time | 4.2 (3.1) | 3.7 (3.3) | 3.9 (3.2)
N2 NREM sleep percentage [Mean (Standard Deviation); unit: percentage of time] — derived from 1-night polysomnography
  percentage of time | 64.2 (10.2) | 62.6 (8.4) | 63.3 (9.2)
N3 NREM sleep percentage [Mean (Standard Deviation); unit: percentage of time] — derived from 1-night polysomnography
  percentage of time | 17.5 (8.8) | 16.4 (7.0) | 16.9 (7.8)
REM sleep percentage [Mean (Standard Deviation); unit: percentage of time] — derived from 1-night polysomnography
  percentage of time | 14.1 (5.5) | 17.0 (7.7) | 15.6 (6.8)
Total sleep time [Mean (Standard Deviation); unit: hours] — derived from 1-night polysomnography
  hours | 5.7 (1.6) | 5.5 (1.6) | 5.6 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Insomnia Severity Index
Description: self reported insomnia symptoms severity by Insomnia severity index . Each item is scored 0 (no problem) - 4 (very big problem) with total between 0-28 (absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).
Time Frame: For BBT-I-first group: on the initial examination (Day 1/Week 1/Month 1), after first treatment course (Day 14/Week 2/Month 1); For zopiclone-first group: after washout period (Day 28/Week 4/Month 1) after second treatment course (Day 42/Week 6/Month 2)
Population: Participants dropped out during the first treatment course and therefore not completed the second treatment course were included only in the analysis for first treatment course and were not analyzed for treatment sequence effect
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BBT-I First Group | Zopiclone First Group
Number analyzed (Participants) | 23 | 19
units on a scale
  Baseline/initial examination | 18.6 (5.2) | 18.9 (3.9)
  First treatment course | 13.1 (5.2) | 14.0 (5.7)
  After washout: number analyzed (Participants) | 23 | 18
  After washout | 14.3 (6.3) | 16.1 (4.7)
  Second treatment course: number analyzed (Participants) | 21 | 18
  Second treatment course | 12.1 (6.1) | 12.8 (5.4)
  After follow-up: number analyzed (Participants) | 18 | 12
  After follow-up | 13.1 (4.7) | 12.7 (5.9)

2. Secondary Outcome: Beck Depression Inventory
Description: 21-item questionnaire assessing (on 4-point Likert scales) the intensity of depressive symptoms in the past week. Minimum score 0, maximum score 63 points. Higher total score represents more severe depressive symptoms
Time Frame: on the initial examination (Day 1/Week 1/Month 1), after first treatment course (Day 14/Week 2/ Month 1), after washout period (Day 28/ Week 4/Month 1), after second treatment course (Day 42/Week 6/Month 8), after second washout (Day 56/Week 8/ Month 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BBT-I First Group | Zopiclone First Group
Number analyzed (Participants) | 23 | 19
units on a scale
  Baseline/initial examination | 11.5 (6.8) | 9.3 (7.3)
  first treatment course | 8.4 (6.8) | 9.4 (8.2)
  After washout: number analyzed (Participants) | 23 | 18
  After washout | 8.4 (8.2) | 9.8 (5.1)
  Second treatment course: number analyzed (Participants) | 23 | 18
  Second treatment course | 9.2 (9.0) | 8.5 (6.2)
  After follow-up: number analyzed (Participants) | 18 | 12
  After follow-up | 9.0 (8.1) | 7.4 (6.2)

3. Secondary Outcome: State Anxiety Subscale (STAI)
Description: State trait anxiety scale is a 2-part questionnaire assessing state (situational) and trait anxiety. State anxiety subscale comprise 20 items rated on a 4-point Likert scale. Minimum score for subscale is 20 and maximum score is 80 points. Higher total score indicates more severe anxiety symptoms
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BBT-I First Group | Zopiclone First Group
Number analyzed (Participants) | 23 | 19
units on a scale
  Baseline/initial examination | 45.1 (8.8) | 43.2 (8.5)
  First treatment course | 43.8 (8.6) | 44.3 (9.1)
  After washout: number analyzed (Participants) | 23 | 18
  After washout | 45.5 (9.0) | 44.5 (9.8)
  Second treatment course: number analyzed (Participants) | 23 | 18
  Second treatment course | 45.1 (9.1) | 44.0 (9.6)
  After follow-up: number analyzed (Participants) | 18 | 12
  After follow-up | 46.9 (6.5) | 44.2 (10.4)

4. Secondary Outcome: Dysfunctional Beliefs About Sleep Scale
Description: questionnaire assessing sleep related cognitions in 16 item rated on a 10-point Likert scale. Minimum score is 0, maximum score is 160 points. Higher total score represents more intensive disfunctional beliefs
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BBT-I First Group | Zopiclone First Group
Number analyzed (Participants) | 23 | 19
units on a scale
  Baseline/initial examination | 105.2 (29.0) | 93.2 (35.0)
  First treatment course | 83.8 (34.8) | 96.4 (36.4)
  After washout: number analyzed (Participants) | 23 | 18
  After washout | 84.76 (36.9) | 103.6 (32.2)
  Second treatment course: number analyzed (Participants) | 23 | 18
  Second treatment course | 84.5 (39.8) | 89.2 (35.4)
  After follow-up: number analyzed (Participants) | 18 | 12
  After follow-up | 62.8 (34.5) | 92.0 (34.5)

5. Secondary Outcome: Sleep Hygiene Index
Description: questionnaire assessing sleep related behavior in 13 item rated on a 5-point Likert scale.Minimum score 13 points and maximum score 65 points. Higher total score represents worse sleep hygiene
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BBT-I First Group | Zopiclone First Group
Number analyzed (Participants) | 23 | 19
units on a scale
  Baseline/initial examination | 26.8 (7.4) | 25.2 (5.9)
  First treatment course | 24.0 (5.6) | 25.0 (6.9)
  After washout: number analyzed (Participants) | 23 | 18
  After washout | 24.7 (6.0) | 25.5 (7.4)
  Second treatment course: number analyzed (Participants) | 23 | 18
  Second treatment course | 24.7 (6.6) | 24.3 (6.6)
  After follow-up: number analyzed (Participants) | 18 | 12
  After follow-up | 23.8 (6.5) | 25.2 (7.6)

6. Secondary Outcome: Pittsburgh Sleep Quality Index
Description: 19-item questionnaire evaluating sleep quality over the past month. The first 4 items are open questions, items 5 to 19 are rated on a 4-point Likert scale. A total score range from 0 to 21. A score > 5 suggests poor sleep quality.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BBT-I First Group | Zopiclone First Group
Number analyzed (Participants) | 23 | 19
units on a scale
  Baseline/initial examination | 13.4 (3.6) | 11.9 (4.1)
  First treatment course | 10.5 (4.5) | 11.3 (4.1)
  After washout: number analyzed (Participants) | 23 | 18
  After washout | 11.3 (4.4) | 12.7 (3.8)
  Second treatment course: number analyzed (Participants) | 23 | 18
  Second treatment course | 10.8 (4.4) | 11.7 (4.8)
  After follow-up: number analyzed (Participants) | 18 | 12
  After follow-up | 11.2 (4.9) | 11.1 (4.7)

7. Secondary Outcome: Trait Anxiety Subscale (STAI)
Description: STAI is a 2-part questionnaire assessing state (situational) and trait anxiety. Trait anxiety subscale comprise 20 items rated on a 4-point Likert scale. Minimum score for each subscale is 20 and maximum score is 80 points. Higher total score indicates more severe anxiety symptoms
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BBT-I First Group | Zopiclone First Group
Number analyzed (Participants) | 23 | 19
units on a scale
  Baseline/initial examination | 48.7 (6.9) | 48.3 (8.1)
  First treatment course | 48.3 (8.1) | 48.3 (8.6)
  After washout: number analyzed (Participants) | 23 | 18
  After washout | 48.6 (7.6) | 49.3 (7.0)
  Second treatment course: number analyzed (Participants) | 23 | 18
  Second treatment course | 46.3 (9.5) | 48.5 (8.3)
  After follow-up: number analyzed (Participants) | 18 | 13
  After follow-up | 46.3 (8.6) | 48.8 (10.7)

8. Other Pre Specified Outcome: Toronto Alexithymia Scale (TAS-20)
Description: Degree of alexithymia evaluated by Toronto Alexithymia scale (20 questions) Measure Description: 0-100 scores. higher values represent worse outcome
Time Frame: once at baseline assessment
Population: All randomised participants who filled baseline set of questionnaires
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Zopiclone First, Then BBT-I | BBT-I First, Then Zopiclone
Number analyzed (Participants) | 19 | 23
scores on a scale | 49.83 (15.9) | 49.33 (10.0)

9. Other Pre Specified Outcome: Sleep Latency
Description: time period from bedding to sleep onset
Time Frame: once at baseline assessment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Zopiclone First, Then BBT-I | BBT-I First, Then Zopiclone
Number analyzed (Participants) | 19 | 23
minutes | 38.53 (21.7) | 54.5 (51.0)

10. Other Pre Specified Outcome: Total Sleep Time
Description: total sleep episode minus wake time
Time Frame: once at baseline assessment
Population: Analysis included all randomized participants
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Zopiclone First, Then BBT-I | BBT-I First, Then Zopiclone
Number analyzed (Participants) | 19 | 23
hours | 5.72 (1.6) | 5.51 (1.6)

11. Other Pre Specified Outcome: Sleep Efficiency
Description: Prercentage of Total Bed Time
Time Frame: once at baseline assessment
Population: Analysis included all participants who were randomized and filled set of questionnaires at baseline assessment
Measure: Mean (Standard Deviation); unit: percentage of polysomnogram time
Arm/Group | Zopiclone First, Then BBT-I | BBT-I First, Then Zopiclone
Number analyzed (Participants) | 19 | 23
percentage of polysomnogram time | 64.68 (17.9) | 63.29 (18.0)

12. Other Pre Specified Outcome: Wake After Sleep Onset
Description: total duration of all periods of wakefulness between sleep onset and final awakening in the morning
Time Frame: once at baseline assessment
Population: All randomised participants who filled baseline set of questionnaires
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Zopiclone First, Then BBT-I | BBT-I First, Then Zopiclone
Number analyzed (Participants) | 19 | 23
minutes | 102.39 (69.0) | 104.75 (76.1)

13. Other Pre Specified Outcome: Amount of Awakenings
Description: Number of awakenings between sleep onset and final morning awakening
Time Frame: once at baseline assessment
Population: All randomised participants who filled baseline set of questionnaires
Measure: Mean (Standard Deviation); unit: awakenings
Arm/Group | Zopiclone First, Then BBT-I | BBT-I First, Then Zopiclone
Number analyzed (Participants) | 19 | 23
awakenings | 13.78 (6.1) | 13.25 (6.9)

14. Other Pre Specified Outcome: N1 NREM Sleep Percentage
Description: Percentage of Total Sleep Time
Time Frame: once at baseline assessment
Population: All randomised participants who filled baseline set of questionnaires
Measure: Mean (Standard Deviation); unit: percentage of total sleep time
Arm/Group | Zopiclone First, Then BBT-I | BBT-I First, Then Zopiclone
Number analyzed (Participants) | 19 | 23
percentage of total sleep time | 4.16 (3.1) | 3.70 (3.3)

15. Other Pre Specified Outcome: N2 NREM Sleep Percentage
Description: Percentage of Total Sleep Time
Time Frame: once at baseline assessment
Population: All randomised participants who filled baseline set of questionnaires
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Zopiclone First, Then BBT-I | BBT-I First, Then Zopiclone
Number analyzed (Participants) | 19 | 23
percentage of time | 64.19 (10.2) | 62.58 (8.4)

16. Other Pre Specified Outcome: N3 NREM Sleep Percentage
Description: Percentage of Total Sleep Time
Time Frame: once at baseline assessment
Population: All randomised participants who filled baseline set of questionnaires
Measure: Mean (Standard Deviation); unit: percentage of total sleep time
Arm/Group | Zopiclone First, Then BBT-I | BBT-I First, Then Zopiclone
Number analyzed (Participants) | 19 | 23
percentage of total sleep time | 17.52 (8.8) | 16.39 (7.0)

17. Other Pre Specified Outcome: REM Sleep Percentage
Description: Percentage of Total Sleep Time
Time Frame: once at baseline assessment
Population: All randomised participants who filled baseline set of questionnaires
Measure: Mean (Standard Deviation); unit: percentage of total sleep time
Arm/Group | Zopiclone First, Then BBT-I | BBT-I First, Then Zopiclone
Number analyzed (Participants) | 19 | 23
percentage of total sleep time | 14.1 (5.5) | 17.0 (7.7)

ADVERSE EVENTS:
Time Frame: 2 months
Description: Adverse effects were evaluated systematically during biweekly visits
Groups:
- BBT-I: Brief behavioral therapy: program included a question-and-answer part; a didactic presentation of sleep regulation mechanisms; the review of causes of onset and chronification of illness; an examination of patient's sleep log; explanation of sleep restriction method and prescription of individual regimen of sleep; explanation of stimulus control method; sleep hygiene education; discussion of relaxation techniques. Participants were supplied with 32 minute audio recording "Relaxation and refreshment session for insomnia" created for this study by Dr. A.Tabidze with verbal relaxing instructions with quiet musical composition behind it. Participants were instructed to listen to this recording in headphones each day for 2-week BBT-I period after laying into bed and turning the light off.
Arm/Group | BBT-I | Zopiclone
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/41
Other Adverse Events (participants affected / at risk) | 0/42 | 2/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BBT-I (N=42) | Zopiclone (N=41)
rash hypersensitivity reaction to zopiclone (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
bitter taste (Hepatobiliary disorders) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-03-18): https://cdn.clinicaltrials.gov/large-docs/83/NCT03339583/Prot_SAP_000.pdf
  • Informed Consent Form (2015-03-18): https://cdn.clinicaltrials.gov/large-docs/83/NCT03339583/ICF_001.pdf